CLINICAL TRIAL: NCT05183269
Title: Virtual Reality for Pain Control During Extracorporeal Shock Wave Lithotripsy: a Prospective, Comparative, Randomized Study at a Single Institution
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: AZ Sint-Lucas Gent (Other)
Responsible Party: Principal Investigator, Luc Merckx, docter, AZ Sint-Lucas Gent
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2018-44
Record Dates: First submitted 2021-12-21; First posted 2022-01-10 (Actual); Last update posted 2022-01-10 (Actual); Status verified 2021-12

CONDITIONS: Stone, Kidney; Stone Ureter
Keywords: Virtual Reality; Shock-wave Lithotripsy; Pain control
MeSH Terms: conditions — Kidney Calculi; Ureterolithiasis; Agnosia

STUDY DESIGN:
Intervention Model Description: Control arm: diclofenac 100 mg suppository + local lidocain/prilocain cream (EMLA 5g, Aspen) Intervention arm: diclofenac 100 mg suppository + local lidocain/prilocain cream (EMLA 5g, Aspen) + Oncomfort virtual reality monitor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual reality (Experimental): Normal procedure with the use of a virtual reality monitor
  Interventions: Device: Oncomfort virtual reality monitor (Oncomfort SA, Wavre, Belgium)
- no virtual reality (No Intervention): Normal procedure without the use of a virtual reality monitor

INTERVENTIONS:
Device: Oncomfort virtual reality monitor (Oncomfort SA, Wavre, Belgium) — Use of the Oncomfort virtual reality monitor
  Arms: Virtual reality

SUMMARY:
The aim of this study is to prospectively analyze patient satisfaction, pain, delivered energy and clinical effectiveness of using VR as a complimentary treatment modality during SWL.

DETAILED DESCRIPTION:
The patients were randomized in two groups SWL with VR and SWL without VR. When a patient was randomized for a VR session we put on the monitor after adequate patient positioning. We used the Oncomfort Sedakit.

The size and location of stone pre-treatment was measured based on the best available imaging tool (CT>RX/ultrasonography) using the maximal stone diameter. The locations of the stones were described as upper pole stones, midpolar stones, lower pole stones, renal pelvis stones and proximal ureteric stones. Each SWL treatment was standardized using diclofenac 100 mg suppository as analgesic and local lidocain/prilocain cream (EMLA 5g, Aspen) to numb the skin. Visualization of the stone was done by fluoroscopy of ultrasonography, as these proved to be equivalent (Van Besien et al. 2017).

A specific and standardized ramping protocol was applied. After finishing this protocol, the energy level could be raised further depending on the level of discomfort of the patient.

Directly after the procedure, the patients were asked to complete a questionnaire where they were asked to write down the experienced amount of pain during the procedure on a VAS of 10 cm and the satisfaction level using a Likert-scale. The total delivered energy was noted.

Two weeks after every SWL session, follow-up imaging (ultrasound and plain abdominal radiography) was performed by a radiologist. Residual stone size was estimated on plain abdominal radiography or ultrasonography. The radiologist was blinded for the randomization process. Practitioner and patient were not. After each SWL the clinical outcome was noted.

ELIGIBILITY:
Inclusion Criteria:

- Patients with renal or ureteric stones in need of a shock-wave lithotripsy. The indication was based on the European association of urology guidelines

Exclusion Criteria:

* none

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 166 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2021-09-13 (Actual); Study Completion 2021-09-13 (Actual)

PRIMARY OUTCOMES:
Pain levels | right after the procedure
  Pain levels determined by a VAS-score

SECONDARY OUTCOMES:
Satisfaction levels | right after the procedure
  Satisfaction levels determined by a LIKERT-scale
Total delivered energy | right after the procedure
  The total delivered energy during the shock-wave lithotripsy
Clinical success | 2 weeks after the procedure
  We defined clinical success as stone-free patients or patients with asymptomatic residual fragments ≤ 4 mm after 1 or more ESWL-sessions

CONTACTS AND LOCATIONS:
Locations (1):
- AZ Sint-Lucas, Ghent, Oost-Vlaanderen, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Weynants L, Chys B, D'hulst P, Merckx L, Van Besien J, Tailly T. Virtual reality for pain control during shock wave lithotripsy: a randomized controlled study. World J Urol. 2023 Feb;41(2):589-594. doi: 10.1007/s00345-023-04280-8. Epub 2023 Jan 21. PMID 36680576